CLINICAL TRIAL: NCT02643797
Title: Medical Assistant Health Coaching for Diabetes in Diverse Primary Care Settings
Acronym: MAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Prinicipal Investigator, Scripps Whittier Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18DK104250-01A1 (NIH)
Record Dates: First submitted 2015-11-30; First posted 2015-12-31 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: diabetes; medical assistant; health coach; glycemic control; pragmatic trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group: MA Health Coaching (Experimental): Patients in the intervention group will receive the "MA Health Coaching" intervention during their primary care visits, as well a follow-up calls to encourage/monitor progress and offer support.
  Interventions: Behavioral: Medical Assistant Health Coaching
- Usual Care (No Intervention): Patients in this group will receive "treatment as usual" during their primary care visits.

INTERVENTIONS:
Behavioral: Medical Assistant Health Coaching — One-on-one behavioral health screening and tailored intervention by the MA health coach with patients who have type 2 diabetes.
  Other Names: MAC
  Arms: Intervention Group: MA Health Coaching

SUMMARY:
This study is a cluster (clinic level) randomized pragmatic trial to compare the effectiveness of MA Health Coaching (MAC) delivered by non-clinician primary care staff (i.e., MAs) versus usual care (UC) in improving diabetes clinical control among individuals with poorly controlled type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
The study will be conducted in the primary care environments of two distinct, yet representative healthcare systems in San Diego County: Neighborhood Healthcare (a San Diego County FQHC system and designated Patient-Centered Medical Home, serving predominantly ethnic minority, low income patients) and Scripps (a large, non-profit, private insurance-based health system, serving predominantly Caucasian, middle-to-higher income patients). Six hundred patients at intervention (n=2; patient N=300) and control (n=2; patient N=300) clinics, aged 18 and older, with T2DM, and glycosylated hemoglobin (HbA1c) ≥ 8.0%, and/or low-density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL, and/or systolic blood pressure (SBP) ≥ 140 within the last 60 days, will be identified and enrolled using electronic health records (EHRs). Primary clinical outcomes of HbA1c, LDL-C, and SBP assessed as part of quarterly (or annual, for LDL-C), standard-of-care medical visits will be extracted from EHRs over 12 months. Changes in patient-reported behavioral (diabetes self-care) and psychosocial (quality of life, patient activation) outcomes will be evaluated via telephone assessment in a subset of intervention and control (N=300 total) participants at baseline, month 6, and month 12. A thorough process evaluation will be conducted to establish reach, acceptability/feasibility, adoption/maintenance, and fidelity of the intervention and will integrate patient, MA, and primary care provider perspectives. Cost-effectiveness will also be examined from the health system perspective. Principles of community engaged research were incorporated in intervention and study planning and will be sustained throughout the research period.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a patient at selected Scripps or Neighborhood Healthcare clinic,
2. Must be age 18 years or older,
3. Must have a T2DM diagnosis,
4. Must show evidence of poor clinical control, defined as HbA1c ≥ 8% and/or LDL-C ≥ 100 mg/dL, and/or SBP ≥ 140 mmHg.

Exclusion Criteria:

None as this is a pragmatic trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-04-19 (Actual)

PRIMARY OUTCOMES:
Glycosylated Hemoglobin (Hba1c); % units | 12 months
Low-density lipoprotein-cholesterol (LDL-c); mg/dL units | 12 months
Systolic blood pressure (SBP); mmHg units | 12 months

SECONDARY OUTCOMES:
Summary of Diabetes Self-Care Activities (SDSCA) - patient-reported outcome | 12 months
Patient Activation Measure (PAM) - patient-reported outcome | 12 months
Patient Reported Outcomes Measurement Information System (PROMIS) General Health Scale - patient-reported outcome | 12 months
Patient Assessment of Care for Chronic Conditions (PACIC) - patient-reported outcome | 12 months
Morisky Medication Adherence Scale (MMAS) - patient-reported outcome | 12 months

OTHER OUTCOMES:
Cost-effectiveness using the United Kingdom Prospective Diabetes Study (UKPDS) Outcomes Model | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Whittier Diabetes Institute; Linda Gallo, PhD, Principal Investigator — San Diego State University
Locations (1):
- Scripps Whittier Diabetes Institute, La Jolla, California, United States